CLINICAL TRIAL: NCT01162603
Title: Comparative Evaluation of Intraocular Pressure During the 24 Hour in Patients Affected by Primary Open-angle Glaucoma and Ocular Hypertension: Latanoprost 0.005% Versus Tafluprost 0.0015% Ophthalmic Solutions
Brief Title: Latanoprost Versus Tafluprost: 24-hour Intraocular Pressure (IOP)
Acronym: SAF-24H-IOP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Collaborators: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Luciano Quaranta, MD, Associate Professor in Ophthalmology, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AOBS-SAF-01
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — tafluprost; Ophthalmic Solutions; Latanoprost

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAFLUPROST 0.0015% EYEDROPS (Experimental): Tafluprost 0.0015% preservative-free ophthalmic solution will be given once a day at the evening,in patients with primary open angle glaucoma (POAG) and/or ocular hypertension (OHT) at first diagnosis. IOP values after three months of treatment will be evaluated throughout the 24-hour by the means of Goldmann and Perkins applanation tonometry.
  Interventions: Device: Goldmann and Perkins applanation tonometry; Drug: TAFLUPROST 0.0015% EYEDROPS
- LATANOPROST 0.005% EYEDROPS (Active Comparator): Latanoprost 0.005% preservative-added ophthalmic solution will be given once a day at the evening,in patients with primary open angle glaucoma (POAG) and/or ocular hypertension (OHT) at first diagnosis. IOP values after three months of treatment will be evaluated throughout the 24-hour by the means Goldmann and Perkins applanation tonometry.
  Interventions: Device: Goldmann and Perkins applanation tonometry; Drug: LATANOPROST 0.005% EYEDROPS

INTERVENTIONS:
Device: Goldmann and Perkins applanation tonometry — IOP values will be assessed by the means of Goldmann or Perkins applanation tonometry at the following time-points: 10AM (± 1 hour), 2PM (± 1 hour), 6PM (± 1 hour), 10PM (± 1 hour), 2AM (± 1 hour) and 6AM (± 1 hour) after three months of treatment
  Other Names: Saflutan, Merck Sharp & Dhome; Latanoprost 0.005% generic drug
Drug: TAFLUPROST 0.0015% EYEDROPS — Tafluprost 0.0015% preservative-free ophthalmic solution
  Other Names: Saflutan, MSD
  Arms: TAFLUPROST 0.0015% EYEDROPS
Drug: LATANOPROST 0.005% EYEDROPS — Latanoprost 0.005% preservative-added ophthalmic solution
  Other Names: Latanoprost 0.005% eyedrops generic drug
  Arms: LATANOPROST 0.005% EYEDROPS

SUMMARY:
* Main objective is to compare the ability of Latanoprost 0.005% preservative-added ophthalmic solution versus Tafluprost 0.0015% preservative-free ophthalmic solution, both given once a day at the evening, in reducing 24-hour intraocular pressure (IOP) in patients with primary open angle glaucoma (POAG) and/or ocular hypertension (OHT) at first diagnosis. First efficacy variable will be the difference between mean nocturnal IOP values after three months of treatment: nocturnal IOP is defined as the mean value between 2AM and 6AM measurements.
* Secondary objectives will be the comparison between Latanoprost 0.005% and Tafluprost 0.0015% ophthalmic solution about:

  * Mean 24-hour IOP values after three months of treatment
  * IOP values at these time-points: 10AM (± 1 hour), 2PM (± 1 hour), 6PM (± 1 hour), 10PM (± 1 hour), 2AM (± 1 hour) and 6AM (± 1 hour) after three months of treatment

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients > 45 years
* Damage of the optic nerve and alterations of the visual field in case of POAG, no defects at the optic nerve and at the visual field in case of OHT
* Untreated IOP > 24 mm Hg but < 32 mm Hg in at least one eye at baseline (10AM) and central corneal thickness between 500 and 600 μm
* Negative pregnancy test (fertile women). Fertile women attending the study must express clear will to avoid pregnancy during all the study period and in the next three months
* Informed consent before starting the study

Exclusion Criteria:

* Secondary glaucoma (Sturge-Weber syndrome, Neurofibromatosis I, neovascular glaucoma, steroid glaucoma, etc)
* Anterior segment anomalies (cataract, irido-corneal disgenesy, congenital ectropion uvae, etc)
* Past ocular surgery, except cataract surgery in the previous 6 months
* Corneal abnormalities that can influence IOP measurements (corneal oedema)
* Positive pregnancy test or breast-feeding woman. No will to avoid pregnancy during all the study period and in the next three months

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure | 24-hour
  Primary endpoint of this crossover trial is to compare the ability of Latanoprost 0.005% preservative-added ophthalmic solution versus Tafluprost 0.0015% preservative-free ophthalmic solution, both given once a day at the evening, in reducing 24-hour intraocular pressure (IOP) in patients with primary open angle glaucoma (POAG) and/or ocular hypertension (OHT) at first diagnosis. First efficacy variable will be the difference between mean nocturnal IOP values after three months of treatment: nocturnal IOP is defined as the mean value between 2AM and 6AM measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Quaranta, MD, Principal Investigator — Università degli Studi di Brescia
Locations (2):
- Glaucoma Unit, 1st University Department of Ophthalmology, Aristotle University, AHEPA Hospital, Thessaloniki, Greece
- USVD "Centro per lo studio del glaucoma" Spedali civili di Brescia, Brescia, Italy

REFERENCES:
- [Background] Kuwayama Y, Komemushi S; Tafluprost Multi-center Study Group. [Intraocular pressure lowering effect of 0.0015% tafluprost as compared to placebo in patients with normal tension glaucoma: randomized, double-blind, multicenter, phase III study]. Nippon Ganka Gakkai Zasshi. 2010 May;114(5):436-43. Japanese. PMID 20545217
- [Background] Uusitalo H, Pillunat LE, Ropo A; Phase III Study Investigators. Efficacy and safety of tafluprost 0.0015% versus latanoprost 0.005% eye drops in open-angle glaucoma and ocular hypertension: 24-month results of a randomized, double-masked phase III study. Acta Ophthalmol. 2010 Feb;88(1):12-9. doi: 10.1111/j.1755-3768.2010.01862.x. PMID 20420586
- [Background] Aihara M. Clinical appraisal of tafluprost in the reduction of elevated intraocular pressure (IOP) in open-angle glaucoma and ocular hypertension. Clin Ophthalmol. 2010 Mar 24;4:163-70. doi: 10.2147/opth.s6368. PMID 20390038
- [Result] Hommer A, Mohammed Ramez O, Burchert M, Kimmich F. IOP-lowering efficacy and tolerability of preservative-free tafluprost 0.0015% among patients with ocular hypertension or glaucoma. Curr Med Res Opin. 2010 Aug;26(8):1905-13. doi: 10.1185/03007995.2010.492030. PMID 20553122
- [Derived] Konstas AG, Quaranta L, Katsanos A, Riva I, Tsai JC, Giannopoulos T, Voudouragkaki IC, Paschalinou E, Floriani I, Haidich AB. Twenty-four hour efficacy with preservative free tafluprost compared with latanoprost in patients with primary open angle glaucoma or ocular hypertension. Br J Ophthalmol. 2013 Dec;97(12):1510-5. doi: 10.1136/bjophthalmol-2012-303026. Epub 2013 May 16. PMID 23681371